CLINICAL TRIAL: NCT05652621
Title: Clinical Efficacy and Mechanism of Probiotics in the Adjuvant Treatment of Ulcerative Colitis and Irritable Bowel Syndrome
Brief Title: Efficacy of Probiotics in Patients With IBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FirstAffiliatedHXinxiangMC
Record Dates: First submitted 2022-09-09; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-07

CONDITIONS: Ulcerative Colitis; Irritable Bowel Syndrome
MeSH Terms: conditions — Colitis, Ulcerative; Irritable Bowel Syndrome | interventions — Probiotics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic intervention group (Experimental): Adjuvant treatment of UC and IBS with "Three-high Probiotics" is given to patients three times a day, one pack of 2g, lasting for 1-4 months.
  Interventions: Dietary Supplement: probiotics

INTERVENTIONS:
Dietary Supplement: probiotics — Resistant dextrin (water-soluble dietary fiber), Lactobacillus reuteri PLBK1, Luo Lactobacillus delbrueckii, Lactobacillus griffii PLBK3, Lactobacillus acidophilus PLBK4, Bifidobacterium lactis PLBK5）

SUMMARY:
This research group plans to take patients with mild to moderate UC and diarrhea IBS diagnosed in the First Affiliated Hospital of Xinxiang Medical College as examples, and divide them into UC group and IBS group; Each group was randomly divided into two groups, namely, conventional treatment+probiotics group and conventional treatment+probiotics placebo group.Starting from the intervention of probiotics on intestinal flora to alleviate intestinal injury caused by UC and IBS patients, the indicators of intestinal flora, serum inflammatory factors, metabolites in vivo, intestinal barrier-related protein expression, and fecal short-chain fatty acid level were detected to explore the clinical efficacy, intestinal protective effect and mechanism of probiotics in adjuvant treatment of UC and IBS patients.To provide new methods and new ideas for refractory UC and IBS, so as to improve the cure rate of UC and IBS, reduce the recurrence rate, relieve the physical and mental pain and economic burden of patients, and provide new ideas for the development and utilization of functional probiotics. It also seeks biosafety evidence for the future use of probiotics in antibiotic environment.

DETAILED DESCRIPTION:
Some studies suggest that IBS is related to UC, and it is speculated that IBS may be a mild UC. Some researchers have also reported that more and more UC patients have irritable bowel syndrome-like symptoms unrelated to intestinal inflammatory activities in remission.At present, it is generally believed that the imbalance of intestinal flora is the main cause of UC and IBS. At present, antibiotics are still the main drugs to treat this disease.Antibiotic treatment often destroys the intestinal microecology, which makes the intestinal microecology unbalanced. Therefore, it is of great guiding significance to find a safe and effective way of dietary intervention.Therefore, our research group induced mice with Dextran Sulfate Sodium Salt (DSS), and successfully established a mouse ulcerative colitis model. On this basis, we used HE staining (histological score), IHC, qPCR and other methods to explore the compound functional mixed strains of probiotics (probiotics for short, The ingredients include: resistant dextrin (water-soluble dietary fiber), Lactobacillus reuteri PLBK1, Lactobacillus reuteri PLBK2, Lactobacillus Grignard PLBK3, Lactobacillus acidophilus PLBK4, Bifidobacterium lactis PLBK5) and their metabolites (feces) to assist the molecular mechanism of ulcerative colitis. The experimental results show that probiotics can significantly improve the symptoms of ulcerative colitis induced by DSS and promote the remission of enteritis.Therefore, in view of the research foundation that our animal experiments have achieved remarkable results, our research group carried out a clinical trial of human medicine in the First Affiliated Hospital of Xinxiang Medical College, and further explored the intervention of probiotics in intestinal flora to assist in the treatment of inflammation. Clinical effect and mechanism of sexual bowel disease. To provide new methods and new ideas for improving the cure rate of UC and IBS, reducing the recurrence rate, alleviating the physical and mental pain and economic burden of patients; At the same time, it provides new ideas for the development and utilization of functional probiotics. It also seeks biosafety evidence for the future use of probiotics in antibiotic environment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ulcerative colitis
* Clinical diagnosis of irritable bowel
* Can swallow probiotic pellets as required

Exclusion Criteria:

* indeterminate colitis,suspected IBD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-31 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of intestinal flora | 4-12 weeks
  collecting the feces of patients before and after taking medicine, and carrying out genomics analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan, China